CLINICAL TRIAL: NCT00392613
Title: RAte Control Efficacy in Permanent Atrial Fibrillation, a Comparison Between Lenient Versus Strict Rate Control in Patients With and Without Heart Failure.
Brief Title: RAte Control Efficacy in Permanent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003B118
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2007-07

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: Strict versus lenient rate control

SUMMARY:
The investigators hypothesis is that in patients with permanent AF lenient rate control is not inferior to strict rate control in terms of cardiovascular mortality, morbidity, neurohormonal activation, NYHA class for heart failure, left ventricular function, left atrial size, quality of life and costs. Lenient rate control is defined as a resting heart rate <110 bpm.Strict rate control is defined as a mean resting heart rate < 80 beats per minute (bpm) and heart rate during minor exercise < 110 bpm. Patients will be seen after 1, 2, 3 months (for titration of rate control drugs) and thereafter yearly.

DETAILED DESCRIPTION:
Study objectives:

1. To show that lenient rate control is not inferior to strict rate control in terms of cardiovascular mortality and morbidity
2. To show that lenient rate control is not inferior to strict rate control in terms of all cause mortality, cardiovascular hospitalizations, NYHA class for exercise tolerance, left ventricular function and left atrial size, quality of life, neurohormonal activation as measured by NT-proBNP, hospitalization for heart failure, syncope, sustained ventricular tachycardia, appropriate shocks or anti-tachycardia pacing of ICD for ventricular arrhythmias, cardiac arrest, and pacemaker implantations, stroke, systemic emboli, and bleeding, unstable angina pectoris and myocardial infarction, costs and renal function

ELIGIBILITY:
Inclusion Criteria:

* Patients with a current episode of permanent AF < 12 months.
* Age </= 80 years.
* Mean resting heart rate > 80 beats per minute with or without rate control medication
* Oral anticoagulation (or aspirin if no risk factors for thromboembolic complications are present).

Exclusion Criteria:

* Paroxysmal AF
* Known contra-indications for either strict or lenient rate control (e.g. previous adverse effects on negative chronotropic drugs).
* Unstable heart failure defined as NYHA IV heart failure and heart failure necessitating hospital admission < 3 months before inclusion.
* Cardiac surgery < 3 months.
* Any stroke.
* Current or foreseen pacemaker and/ or cardiac resynchronization therapy.
* Signs of sick sinus syndrome or AV conduction disturbances (i.e. symptomatic bradycardia or asystole > 3 seconds or escape rate < 40 beats per minute in awake symptom-free patients).
* Untreated hyperthyroidism or < 3 months euthyroidism.
* Inability to walk or bike.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality
Heart failure
Stroke
Bleeding
Syncope
Ventricular tachycardia
PM / ICD implantation
Cardiac arrest
Life-threatening adverse effects of RC drugs

SECONDARY OUTCOMES:
All cause mortality
All cause hospitalizations
Exercise tolerance
LV function and left atrial size
Quality of life
NT-proBNP
Costs
Renal function

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C Van Gelder, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Groenveld HF, Crijns HJ, Van den Berg MP, Van Sonderen E, Alings AM, Tijssen JG, Hillege HL, Tuininga YS, Van Veldhuisen DJ, Ranchor AV, Van Gelder IC; RACE II Investigators. The effect of rate control on quality of life in patients with permanent atrial fibrillation: data from the RACE II (Rate Control Efficacy in Permanent Atrial Fibrillation II) study. J Am Coll Cardiol. 2011 Oct 18;58(17):1795-803. doi: 10.1016/j.jacc.2011.06.055. PMID 21996393
- [Derived] Smit MD, Crijns HJ, Tijssen JG, Hillege HL, Alings M, Tuininga YS, Groenveld HF, Van den Berg MP, Van Veldhuisen DJ, Van Gelder IC; RACE II Investigators. Effect of lenient versus strict rate control on cardiac remodeling in patients with atrial fibrillation data of the RACE II (RAte Control Efficacy in permanent atrial fibrillation II) study. J Am Coll Cardiol. 2011 Aug 23;58(9):942-9. doi: 10.1016/j.jacc.2011.04.030. PMID 21851883
- [Derived] Van Gelder IC, Groenveld HF, Crijns HJ, Tuininga YS, Tijssen JG, Alings AM, Hillege HL, Bergsma-Kadijk JA, Cornel JH, Kamp O, Tukkie R, Bosker HA, Van Veldhuisen DJ, Van den Berg MP; RACE II Investigators. Lenient versus strict rate control in patients with atrial fibrillation. N Engl J Med. 2010 Apr 15;362(15):1363-73. doi: 10.1056/NEJMoa1001337. Epub 2010 Mar 15. PMID 20231232